CLINICAL TRIAL: NCT02057159
Title: A Phase II Study of NeuroVax™, a Therapeutic TCR Peptide Vaccine for SPMS of Multiple Sclerosis
Brief Title: A Study of NeuroVax™, a Therapeutic TCR Peptide Vaccine for SPMS of Multiple Sclerosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immune Response BioPharma, Inc. (Industry)
Collaborators: cro (Ambiguous)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IR902-231
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Secondary Progress Multiple Sclerosis; Multiple Sclerosis
Keywords: Secondary Progress Multiple Sclerosis; SPMS; Multiple Sclerosis; NeuroVax
MeSH Terms: conditions — Multiple Sclerosis | interventions — NeuroVax vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NeuroVax (Experimental): NeuroVax
  Interventions: Biological: NeuroVax
- IFA Placebo (Placebo Comparator): IFA Placebo
  Interventions: Biological: IFA Placebo

INTERVENTIONS:
Biological: NeuroVax — TCR peptides in IFA
  Arms: NeuroVax
Biological: IFA Placebo — IFA Placebo
  Arms: IFA Placebo

SUMMARY:
Multi-center, randomized , double-blind, placebo-controlled , two arm parallel design study of NeuroVax™ vs. Incomplete Freund's Adjuvant ( I F A) placebo. 200 subjects with Secondary Progressive SPMS

DETAILED DESCRIPTION:
Objectives:The primary objective is to compare between treatment groups the cumulative number of new gadolinium enhancing (Gd+) lesions on brain MRI at weeks 24, 32, 40 and 48 i n subjects with secondary progressive MS. Secondary objectives include additional MRI measurements, analyses of clinical relapses, measures of neurologic disability, immunologic evaluations, and safety.

Study Design: Multi-center, randomized , double-blind, placebo-controlled , two arm parallel design study of NeuroVax™ vs. Incomplete Freund's Adjuvant ( I F A) placebo.

Subject Population: 200 subjects with Secondary Progressive SPMS MS, with an EDSS score >= 3.5 , and meeting all inclusion/exclusion criteria, will be enroll in this study. Subjects will be randomized equally to NeuroVax™ or I F A

,1 0 0 per arm .

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 and 50 years of age, inclusive.
* Definite MS by the revised McDonald criteria (2005) (Appendix A), with a Secondary Progressive course.
* Expanded Disability Status Scale (EDSS) >=score 3.5 (Appendix B).
* Two or more documented clinical relapses of MS in the preceding 24 months OR one documented clinical relapse of MS in the preceding 1 2 months prior to screening .
* Laboratory values within the following limits:

  * Creatinine 1 . 5 x high normal.
  * Hemoglobin

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2023-03-09 (Estimated); Study Completion 2023-03-09 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare between treatment groups the cumulative number of new gadolinium enhancing (Gd+) lesions on brain MRI at up to 48 weeks in subjects with secondary progressive MS | up to 48 weeks

SECONDARY OUTCOMES:
Secondary MRI measurements objectives include additional MRI measurements, analyses of clinical relapses, measures of neurologic disability, immunologic evaluations, and safety. | 48 Weeks
  Secondary MRI measurements
Analyses of clinical relapses | 48 Weeks
  Analyses of clinical relapses
Measures of neurologic disability EDSS score | 48 Weeks
  Measures of neurologic disability EDSS score
Immunologic evaluations | 48 Weeks
  Immunologic evaluations
Safety Evaluation | 48 Weeks
  Safety Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bartholomew, Ph.D, Study Director — Immune Response BioPharma, Inc.
Locations (1):
- CRO, San Diego, California, United States